CLINICAL TRIAL: NCT02318290
Title: Opioids Withdrawal Syndrome in Critically Ill Patients: a Multicenter Prospective Cohort Study
Acronym: WAAICUP
Status: Completed | Type: Observational
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, David Williamson, Full Clinical Professor, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Other Study IDs: 2014-1112
Record Dates: First submitted 2014-12-09; First posted 2014-12-17 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Substance Withdrawal Syndrome
Keywords: Analgesia; Critical Care; Hypnotics and Sedatives
MeSH Terms: conditions — Substance Withdrawal Syndrome; Agnosia | interventions — Opiate Alkaloids; Analgesics; Narcotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critically ill patients: Mechanically ventilated critically ill patients receiveing opiates for more than 96 hours will be prospectively followed for the emergence of withdrawal symptoms upon weaning of opiates
  Interventions: Drug: Opiates

INTERVENTIONS:
Drug: Opiates — Mechanically ventilated patients receiving opiates for more than 96 hours will be evaluated for withdrawal symptoms upon weaning of the opiates
  Other Names: Analgesics; Narcotics

SUMMARY:
Critically ill patients who are mechanically ventilated may require prolonged administration of sedatives and analgesics. Their prolonged use has been associated with withdrawal symptoms upon rapid weaning in critically ill patients. These withdrawal symptoms may be associated with adverse clinical outcomes. Although well studied in the paediatric population, little is known about the epidemiology, risk factors and optimal screening methods in adults. Studying this problem is essential as we strive to develop proper weaning strategies.

Methods: Prospective observational two-center study in critically ill adult patients Objectives: 1) Describe the incidence of iatrogenic withdrawal of sedatives and analgesics in critically ill adult patients and 2) Evaluate the performance of screening tools assessing withdrawal that were developed for the paediatric patient in the adult population.

DETAILED DESCRIPTION:
The objectives of the study are: 1) to describe the incidence of iatrogenic withdrawal of sedatives and analgesics in critically ill adult patients and; 2) Validate screening tools for withdrawal in the adult population.

Hypothesis

1. Symptoms of iatrogenic benzodiazepines and opioids withdrawal occur commonly in mechanically ventilated patients exposed to high doses and/or prolonged infusions and who are rapidly weaned from these therapies.
2. The scales for benzodiazepine and narcotic withdrawal detection used in paediatrics population correlate well with the DSM V diagnosis of withdrawal in an adult ICU population
3. Major risk factors for withdrawal symptoms include longer duration of therapy and higher doses and admission for a medical condition (MICU)

Methods

A prospective multicenter observational study will be carried out in two University-affiliated hospital intensive care units (Hôpital du Sacré-Coeur and Montreal General Hospital). All mechanically ventilated ICU patients receiving continuous infusions of benzodiazepines and/or opioids for more than 96 hours will be prospectively screened daily for withdrawal symptoms by an intensivist. Withdrawal symptoms for opioid and benzodiazepines will be identified using the DSM-V criteria. Patients with moderate to severe head trauma, a severe neurological disease, or prior to admission substance abuse (significant alcohol, illicit or prescription drugs) will be excluded. We will also exclude patients with a regularly prescribed chronic opioid or benzodiazepine use prior to ICU admission. Risk factors for withdrawal including type of agents exposed, dosing, duration of exposure, weaning of agents, organ dysfunction, age, gender, smoking, severity of disease and admission diagnosis will be prospectively collected. The Withdrawal Assessment Tool-1 (WAT-1), a screening tools validated in the paediatric population, will also be administered daily. The criterion validity of this screening tool will be compared to the DSM-V criteria.

ELIGIBILITY:
Inclusion Criteria:

* intermittent use or continuous infusion opioids for at least 96 hours

Exclusion Criteria:

* Patient and/or relatives unable to communicate in French or English
* Patients unable to communicate (consent form and evaluation)
* Patient deaf without appropriate hearing aid
* Patients unable to communicate (consent form and evaluation)
* Imminent and predictable death according to medical team
* Severe brain injury, defined as Glasgow Coma Scale (GCS) score of 8 or less at ICU admission
* Moderate brain injury, defined as GCS between 9 and 12, with elevated intracranial pressure (ICP > 20 mm Hg) who requires ICP monitoring and osmotherapy
* Major confounding factors for withdrawal syndrome by causing shivering, sympathetic drive and autonomic disorders
* Underlying active neurological condition (status epilepticus, encephalopathy, hypoxia)
* Neurological problems are covariates, which would make the assessment of sedation or IWS difficult Patient previously included in the study at any of the two hospitals (readmission to the ICU at a later date during the period of recruitment for the study, limiting to 1 weaning episode per patient)
* Thoracic and cervical spinal cord injury
* Adrenergic response to pain will be difficult to assess
* Unable to assess validated tool: DSM-V, RASS, CAM-ICU
* Narcotic
* If the underlying neurological condition resolves within the 96 hours, the patient may be included in the study
* Substance abuse prior to ICU admission (28)
* Chronic alcohol use defined as alcohol consumption of more than 2 drinks per day and/or more than 14 drinks per week for men and 9 drinks per week for woman as reported by family or as per patient's medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under mechanical ventilation and receiving regular intermittent use or continuous infusion opioids for at least 96 hours
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Opiate withdrawal according to DSM V critieria | From ICU admission to 48 hours post-extubation or a maximum of 14 days passed since the beginning of the initial weaning process
  Opiate withdrawal as evaluated by an intensivist using DSM V criteria

CONTACTS AND LOCATIONS:
Overall Officials: David Williamson, Ph.D., Principal Investigator — Hopital du Sacre-Coeur de Montréal; Marc Perreaut, Pharm.D., Principal Investigator — Montreal General Hospital; Anne Julie Frenette, M.Sc., Principal Investigator — Hopital du Sacre-Coeur de Montréal
Locations (1):
- Hôpital du Sacré-Coeur, Montreal, Quebec, Canada

REFERENCES:
- [Background] Cammarano WB, Pittet JF, Weitz S, Schlobohm RM, Marks JD. Acute withdrawal syndrome related to the administration of analgesic and sedative medications in adult intensive care unit patients. Crit Care Med. 1998 Apr;26(4):676-84. doi: 10.1097/00003246-199804000-00015. PMID 9559604
- [Background] Franck LS, Harris SK, Soetenga DJ, Amling JK, Curley MA. The Withdrawal Assessment Tool-1 (WAT-1): an assessment instrument for monitoring opioid and benzodiazepine withdrawal symptoms in pediatric patients. Pediatr Crit Care Med. 2008 Nov;9(6):573-80. doi: 10.1097/PCC.0b013e31818c8328. PMID 18838937